CLINICAL TRIAL: NCT03210766
Title: Nabilone and THC/CBD for the Treatment of FBSS Refractory Pain
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Principal Investigator, Gioacchino Calapai, Full Professor of Pharmacology, Azienda Ospedaliera Universitaria Policlinico "G. Martino"
Other Study IDs: CAN 01
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: FBSS
Keywords: Cannabinoids, nabilone, FBSS, THC/CBD, refractory pain
MeSH Terms: conditions — Failed Back Surgery Syndrome; Pain, Intractable | interventions — nabilone; Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nabilone: Patients affected by Failed Back Surgery Syndrome (FBSS)
  Interventions: Drug: Nabilone
- THC/CBD: Patients affected by Failed Back Surgery Syndrome (FBSS)
  Interventions: Drug: THC/CBD

INTERVENTIONS:
Drug: Nabilone
  Other Names: Spinal Cord Stimulation
  Groups: Nabilone
Drug: THC/CBD
  Other Names: Spinal Cord Stimulation
  Groups: THC/CBD

SUMMARY:
The aim of this study is to evaluate the efficacy of oral administration of nabilone or THC/CBD administration in combination with spinal cord stimulation (SCS) in FBSS patients refractory to other available therapeutic strategies.

DETAILED DESCRIPTION:
Failed Back Surgery Syndrome (FBSS) is defined as: spinal pain of unknown origin either persisting despite surgical intervention or appearing after surgical intervention for spinal pain originally in the same topographical location.

Several conditions have been identified as causes of FBSS: epidural fibrosis, canal stenosis (global or lateral), foraminal stenosis, retained disc fragment, recurrent disc herniation or degeneration, spinal instability, facet joint pain, sacroiliac joint pain, discitis, adhesive arachnoiditis and others.

Can involve 20% to 40% of patients who have undergone lumbar spine surgery and 0.02% to 2% of the general population suffer from this syndrome.

In FBSS symptoms are the persistence of low back pain, deterioration or recurrence of radiculopathy, sensory and/or motor deficit, sphincter dysfunction.

Chronic opioid therapy does not improve long-term pain management. Similar issues can occur with conservative measures like peridural injections of steroids, intrathecal analgesic infusion and local anesthetics injections. Despite a large part of FBSS patients benefit of radio-frequency treatment and/or spinal cord stimulation (SCS), a small percentage of them doesn't report benefits.

Pain could be treated by drugs modulating endocannabinoid system and it could represent a pharmacological option in a multimodal treatment approach for neuropathic pain.

Authors present a retrospective case series documenting the efficacy and safety of oral administration of cannabinoids agonists (THC/CBD and nabilone) in 20 FBSS patients, presenting moderate to severe chronic pain that not responding to other treatment regimens.

Cannabinoids agonists were administered in association with the practice of spinal cord stimulation (SCS).

Other analgesic therapies were discontinued before the beginning of the treatment.

The study was performed during the period between September 2014 and January 2016 and the duration was up to 12 months.

Characteristics and severity of neuropathic pain were measured using the Douleur Neuropathique 4 questionnaire. The Brief Pain Inventory allows patients to rate the severity of their pain and the degree to which pain interferes with common dimensions of feeling and function.

Patients aged between 45 and 69. All patients received a fixed dose of cannabinoid agonists: treatment was initiated with nabilone 1mg/day or an oleic suspension for oral administration of THC/CBD 25mg/day.

The basal dose was increased depending on effects on pain control. Adverse reactions were treated by decreasing the subscripted dose. If adverse events required the suspension of the administration of the initially prescribed drug, the same was switched with the other available in the study.

ELIGIBILITY:
Inclusion Criteria:

* FBSS with refractory pain
* DN-4 score of 4 or +

Exclusion Criteria:

* Adverse Drug Reaction
* Subject suffers from FBSS that could not quit the previous pharmacological therapy

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that comes to the pain unit, suffer from FBSS refractory pain
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | 2015/1 to 2016/1
  The Brief Pain Inventory allows patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function. BPI has been shown to be an appropriate measure for pain caused by a wide range of clinical conditions. The BPI is an 11-item questionnaire that consists of four 0- to-10 numeric rating scale (NRS) items asking patients to rate their pain at its "worst in the last 24-hours," least in the last 24-hours," "average," and "now," with a 0 indicating "no pain" and 10 representing "pain as bad as you could imagine." The remaining seven BPI items probe the degree to which pain interferes with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life, again using a 0-to-10 value scale. For these interference items, 0 represents "does not interfere" and 10 indicates "interferes completely."
Douleur Neuropathique-4 (DN-4) | 2015/1 to 2016/1
  The DN4 questionnaire consists of a total of 10 items: 7 items related to the characteristics of pain (burning, painful cold, electric shocks) and its association with abnormal sensations (tingling, pins and needles, numbness, itching), and 3 related to neurological examination in the painful area (touch hypesthesia, pinprick hypesthesia, tactile allodynia). The value of 1 was given to each positive item, and 0 value to each negative item. The total score was calculated as the sum of all 10 items and the cutoff value for the diagnosis of neuropathic pain is established as a total score of 4/10.

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Quattrone, MD, Principal Investigator — S. Vincenzo Hospital ASP Messina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burton CV, Kirkaldy-Willis WH, Yong-Hing K, Heithoff KB. Causes of failure of surgery on the lumbar spine. Clin Orthop Relat Res. 1981 Jun;(157):191-9. PMID 7249453
- [Background] Waguespack A, Schofferman J, Slosar P, Reynolds J. Etiology of long-term failures of lumbar spine surgery. Pain Med. 2002 Mar;3(1):18-22. doi: 10.1046/j.1526-4637.2002.02007.x. PMID 15102214
- [Background] Slipman CW, Shin CH, Patel RK, Isaac Z, Huston CW, Lipetz JS, Lenrow DA, Braverman DL, Vresilovic EJ Jr. Etiologies of failed back surgery syndrome. Pain Med. 2002 Sep;3(3):200-14; discussion 214-7. doi: 10.1046/j.1526-4637.2002.02033.x. PMID 15099254
- [Background] Krishna M, Pollock RD, Bhatia C. Incidence, etiology, classification, and management of neuralgia after posterior lumbar interbody fusion surgery in 226 patients. Spine J. 2008 Mar-Apr;8(2):374-9. doi: 10.1016/j.spinee.2006.09.004. Epub 2006 Dec 22. PMID 17433779
- [Background] Hussain A, Erdek M. Interventional pain management for failed back surgery syndrome. Pain Pract. 2014 Jan;14(1):64-78. doi: 10.1111/papr.12035. Epub 2013 Feb 3. PMID 23374545
- [Background] Choi HS, Chi EH, Kim MR, Jung J, Lee J, Shin JS, Ha IH. Demographic characteristics and medical service use of failed back surgery syndrome patients at an integrated treatment hospital focusing on complementary and alternative medicine: a retrospective review of electronic medical records. Evid Based Complement Alternat Med. 2014;2014:714389. doi: 10.1155/2014/714389. Epub 2014 Nov 4. PMID 25530787
- [Background] Shapiro CM. The failed back surgery syndrome: pitfalls surrounding evaluation and treatment. Phys Med Rehabil Clin N Am. 2014 May;25(2):319-40. doi: 10.1016/j.pmr.2014.01.014. PMID 24787336
- [Background] Thomson S. Failed back surgery syndrome - definition, epidemiology and demographics. Br J Pain. 2013 Feb;7(1):56-9. doi: 10.1177/2049463713479096. PMID 26516498
- [Background] Peul WC, van Houwelingen HC, van den Hout WB, Brand R, Eekhof JA, Tans JT, Thomeer RT, Koes BW; Leiden-The Hague Spine Intervention Prognostic Study Group. Surgery versus prolonged conservative treatment for sciatica. N Engl J Med. 2007 May 31;356(22):2245-56. doi: 10.1056/NEJMoa064039. PMID 17538084
- [Background] Chan CW, Peng P. Failed back surgery syndrome. Pain Med. 2011 Apr;12(4):577-606. doi: 10.1111/j.1526-4637.2011.01089.x. Epub 2011 Apr 4. PMID 21463472
- [Background] Khosravi MB, Azemati S, Sahmeddini MA. Gabapentin versus naproxen in the management of failed back surgery syndrome; a randomized controlled trial. Acta Anaesthesiol Belg. 2014;65(1):31-7. PMID 24988825
- [Background] Zencirci B. Analgesic efficacy of oral gabapentin added to standard epidural corticosteroids in patients with failed back surgery. Clin Pharmacol. 2010;2:207-11. doi: 10.2147/CPAA.S12126. Epub 2010 Sep 30. PMID 22291506
- [Background] Abeloos L, De Witte O, Riquet R, Tuna T, Mathieu N. [Long-term outcome of patients treated with spinal cord stimulation for therapeutically refractory failed back surgery syndrome: a retrospective study]. Neurochirurgie. 2011 Jul;57(3):114-9. doi: 10.1016/j.neuchi.2011.07.001. Epub 2011 Sep 9. French. PMID 21907361
- [Background] Van Buyten JP, Al-Kaisy A, Smet I, Palmisani S, Smith T. High-frequency spinal cord stimulation for the treatment of chronic back pain patients: results of a prospective multicenter European clinical study. Neuromodulation. 2013 Jan-Feb;16(1):59-65; discussion 65-6. doi: 10.1111/ner.12006. Epub 2012 Nov 30. PMID 23199157
- [Background] North RB, Kidd D, Shipley J, Taylor RS. Spinal cord stimulation versus reoperation for failed back surgery syndrome: a cost effectiveness and cost utility analysis based on a randomized, controlled trial. Neurosurgery. 2007 Aug;61(2):361-8; discussion 368-9. doi: 10.1227/01.NEU.0000255522.42579.EA. PMID 17762749
- [Background] Sciubba DM, Gokaslan ZL. Spinal cord stimulation for failed back surgery syndrome--does it work and is it cost-effective? Nat Clin Pract Neurol. 2008 Sep;4(9):472-3. doi: 10.1038/ncpneuro0865. Epub 2008 Jul 22. PMID 18648348
- [Background] Boswell MV, Hansen HC, Trescot AM, Hirsch JA. Epidural steroids in the management of chronic spinal pain and radiculopathy. Pain Physician. 2003 Jul;6(3):319-34. PMID 16880879
- [Background] Kim SB, Lee KW, Lee JH, Kim MA, An BW. The effect of hyaluronidase in interlaminar lumbar epidural injection for failed back surgery syndrome. Ann Rehabil Med. 2012 Aug;36(4):466-73. doi: 10.5535/arm.2012.36.4.466. Epub 2012 Aug 27. PMID 22977771
- [Background] Kumar K, Hunter G, Demeria DD. Treatment of chronic pain by using intrathecal drug therapy compared with conventional pain therapies: a cost-effectiveness analysis. J Neurosurg. 2002 Oct;97(4):803-10. doi: 10.3171/jns.2002.97.4.0803. PMID 12405366
- [Background] Tomycz ND, Ortiz V, Moossy JJ. Simultaneous intrathecal opioid pump and spinal cord stimulation for pain management: analysis of 11 patients with failed back surgery syndrome. J Pain Palliat Care Pharmacother. 2010 Dec;24(4):374-83. doi: 10.3109/15360288.2010.523066. PMID 21133746
- [Background] Wong CB, Chen WJ, Chen LH, Niu CC, Lai PL. Clinical outcomes of revision lumbar spinal surgery: 124 patients with a minimum of two years of follow-up. Chang Gung Med J. 2002 Mar;25(3):175-82. PMID 12022738
- [Background] Duggal N, Mendiondo I, Pares HR, Jhawar BS, Das K, Kenny KJ, Dickman CA. Anterior lumbar interbody fusion for treatment of failed back surgery syndrome: an outcome analysis. Neurosurgery. 2004 Mar;54(3):636-43; discussion 643-4. doi: 10.1227/01.neu.0000108423.87889.9e. PMID 15028138
- [Background] Kat'uch V, Pataky F, Kat'uchova J, Gajdos M, Radonak J. [Surgical management of the failed back surgery syndrome (FBSS) using posterior lumbar interbody fusion (PLIF) with posterior transpedicular stabilization]. Rozhl Chir. 2010 Aug;89(7):450-8. Slovak. PMID 20925263
- [Background] Simon A, Seizeur R, Person H, Forlodou P, Dam Hieu P, Besson G. [Anterior lumbar interbody fusion for treatment of failed back surgery syndrome: a retrospective study of 46 cases]. Neurochirurgie. 2009 Jun;55(3):309-13. doi: 10.1016/j.neuchi.2008.09.003. Epub 2008 Dec 16. French. PMID 19091357
- [Background] Esmer G, Blum J, Rulf J, Pier J. Mindfulness-based stress reduction for failed back surgery syndrome: a randomized controlled trial. J Am Osteopath Assoc. 2010 Nov;110(11):646-52. PMID 21135196
- [Background] Manniche C, Asmussen K, Lauritsen B, Vinterberg H, Karbo H, Abildstrup S, Fischer-Nielsen K, Krebs R, Ibsen K. Intensive dynamic back exercises with or without hyperextension in chronic back pain after surgery for lumbar disc protrusion. A clinical trial. Spine (Phila Pa 1976). 1993 Apr;18(5):560-7. doi: 10.1097/00007632-199304000-00007. PMID 8484146
- [Background] Katz JA, Swerdloff MA, Brass SD, Argoff CE, Markman J, Backonja M, Katz N. Opioids for chronic noncancer pain: A position paper of the American Academy of Neurology. Neurology. 2015 Apr 7;84(14):1503-4. doi: 10.1212/WNL.0000000000001485. No abstract available. PMID 25846999
- [Background] Lynch ME, Campbell F. Cannabinoids for treatment of chronic non-cancer pain; a systematic review of randomized trials. Br J Clin Pharmacol. 2011 Nov;72(5):735-44. doi: 10.1111/j.1365-2125.2011.03970.x. PMID 21426373
- [Background] Torrance N, Smith BH, Bennett MI, Lee AJ. The epidemiology of chronic pain of predominantly neuropathic origin. Results from a general population survey. J Pain. 2006 Apr;7(4):281-9. doi: 10.1016/j.jpain.2005.11.008. PMID 16618472
- [Background] Attal N, Bouhassira D. Pharmacotherapy of neuropathic pain: which drugs, which treatment algorithms? Pain. 2015 Apr;156 Suppl 1:S104-S114. doi: 10.1097/01.j.pain.0000460358.01998.15. PMID 25789426
- [Background] Baron R, Binder A, Wasner G. Neuropathic pain: diagnosis, pathophysiological mechanisms, and treatment. Lancet Neurol. 2010 Aug;9(8):807-19. doi: 10.1016/S1474-4422(10)70143-5. PMID 20650402
- [Background] Maier C, Baron R, Sommer C. [Neuropathic pain. How to open the blackbox]. Schmerz. 2015 Oct;29(5):479-80, 482-5. doi: 10.1007/s00482-015-0028-y. German. PMID 26264897
- [Background] Baber Z, Erdek MA. Failed back surgery syndrome: current perspectives. J Pain Res. 2016 Nov 7;9:979-987. doi: 10.2147/JPR.S92776. eCollection 2016. PMID 27853391
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Background] Finnerup NB, Sindrup SH, Jensen TS. The evidence for pharmacological treatment of neuropathic pain. Pain. 2010 Sep;150(3):573-581. doi: 10.1016/j.pain.2010.06.019. PMID 20705215
- [Background] O'Connor AB, Dworkin RH. Treatment of neuropathic pain: an overview of recent guidelines. Am J Med. 2009 Oct;122(10 Suppl):S22-32. doi: 10.1016/j.amjmed.2009.04.007. PMID 19801049
- [Background] Lynch ME, Ware MA. Cannabinoids for the Treatment of Chronic Non-Cancer Pain: An Updated Systematic Review of Randomized Controlled Trials. J Neuroimmune Pharmacol. 2015 Jun;10(2):293-301. doi: 10.1007/s11481-015-9600-6. Epub 2015 Mar 22. PMID 25796592
- [Background] Tsang CC, Giudice MG. Nabilone for the Management of Pain. Pharmacotherapy. 2016 Mar;36(3):273-86. doi: 10.1002/phar.1709. Epub 2016 Feb 29. PMID 26923810
- [Background] Atkinson TM, Rosenfeld BD, Sit L, Mendoza TR, Fruscione M, Lavene D, Shaw M, Li Y, Hay J, Cleeland CS, Scher HI, Breitbart WS, Basch E. Using confirmatory factor analysis to evaluate construct validity of the Brief Pain Inventory (BPI). J Pain Symptom Manage. 2011 Mar;41(3):558-65. doi: 10.1016/j.jpainsymman.2010.05.008. Epub 2010 Dec 4. PMID 21131166
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Ware MA, Doyle CR, Woods R, Lynch ME, Clark AJ. Cannabis use for chronic non-cancer pain: results of a prospective survey. Pain. 2003 Mar;102(1-2):211-6. doi: 10.1016/s0304-3959(02)00400-1. PMID 12620613
- [Background] Pertwee RG. Targeting the endocannabinoid system with cannabinoid receptor agonists: pharmacological strategies and therapeutic possibilities. Philos Trans R Soc Lond B Biol Sci. 2012 Dec 5;367(1607):3353-63. doi: 10.1098/rstb.2011.0381. PMID 23108552
- [Background] Stout SM, Cimino NM. Exogenous cannabinoids as substrates, inhibitors, and inducers of human drug metabolizing enzymes: a systematic review. Drug Metab Rev. 2014 Feb;46(1):86-95. doi: 10.3109/03602532.2013.849268. Epub 2013 Oct 25. PMID 24160757
- [Background] Zuardi AW, Shirakawa I, Finkelfarb E, Karniol IG. Action of cannabidiol on the anxiety and other effects produced by delta 9-THC in normal subjects. Psychopharmacology (Berl). 1982;76(3):245-50. doi: 10.1007/BF00432554. PMID 6285406
- [Background] Booz GW. Cannabidiol as an emergent therapeutic strategy for lessening the impact of inflammation on oxidative stress. Free Radic Biol Med. 2011 Sep 1;51(5):1054-61. doi: 10.1016/j.freeradbiomed.2011.01.007. Epub 2011 Jan 14. PMID 21238581
- [Background] Fernandez-Ruiz J, Sagredo O, Pazos MR, Garcia C, Pertwee R, Mechoulam R, Martinez-Orgado J. Cannabidiol for neurodegenerative disorders: important new clinical applications for this phytocannabinoid? Br J Clin Pharmacol. 2013 Feb;75(2):323-33. doi: 10.1111/j.1365-2125.2012.04341.x. PMID 22625422
- [Background] Izzo AA, Borrelli F, Capasso R, Di Marzo V, Mechoulam R. Non-psychotropic plant cannabinoids: new therapeutic opportunities from an ancient herb. Trends Pharmacol Sci. 2009 Oct;30(10):515-27. doi: 10.1016/j.tips.2009.07.006. Epub 2009 Sep 2. PMID 19729208
- [Background] Hayakawa K, Mishima K, Hazekawa M, Sano K, Irie K, Orito K, Egawa T, Kitamura Y, Uchida N, Nishimura R, Egashira N, Iwasaki K, Fujiwara M. Cannabidiol potentiates pharmacological effects of Delta(9)-tetrahydrocannabinol via CB(1) receptor-dependent mechanism. Brain Res. 2008 Jan 10;1188:157-64. doi: 10.1016/j.brainres.2007.09.090. Epub 2007 Oct 12. PMID 18021759
- [Background] Casarotto PC, Gomes FV, Resstel LB, Guimaraes FS. Cannabidiol inhibitory effect on marble-burying behaviour: involvement of CB1 receptors. Behav Pharmacol. 2010 Jul;21(4):353-8. doi: 10.1097/fbp.0b013e32833b33c5. PMID 20695034
- [Background] Ryberg E, Larsson N, Sjogren S, Hjorth S, Hermansson NO, Leonova J, Elebring T, Nilsson K, Drmota T, Greasley PJ. The orphan receptor GPR55 is a novel cannabinoid receptor. Br J Pharmacol. 2007 Dec;152(7):1092-101. doi: 10.1038/sj.bjp.0707460. Epub 2007 Sep 17. PMID 17876302
- [Background] Russo EB, Burnett A, Hall B, Parker KK. Agonistic properties of cannabidiol at 5-HT1a receptors. Neurochem Res. 2005 Aug;30(8):1037-43. doi: 10.1007/s11064-005-6978-1. PMID 16258853
- [Background] Pazos MR, Mohammed N, Lafuente H, Santos M, Martinez-Pinilla E, Moreno E, Valdizan E, Romero J, Pazos A, Franco R, Hillard CJ, Alvarez FJ, Martinez-Orgado J. Mechanisms of cannabidiol neuroprotection in hypoxic-ischemic newborn pigs: role of 5HT(1A) and CB2 receptors. Neuropharmacology. 2013 Aug;71:282-91. doi: 10.1016/j.neuropharm.2013.03.027. Epub 2013 Apr 12. PMID 23587650
- [Background] Kathmann M, Flau K, Redmer A, Trankle C, Schlicker E. Cannabidiol is an allosteric modulator at mu- and delta-opioid receptors. Naunyn Schmiedebergs Arch Pharmacol. 2006 Feb;372(5):354-61. doi: 10.1007/s00210-006-0033-x. Epub 2006 Feb 18. PMID 16489449
- [Background] Esposito G, Scuderi C, Valenza M, Togna GI, Latina V, De Filippis D, Cipriano M, Carratu MR, Iuvone T, Steardo L. Cannabidiol reduces Abeta-induced neuroinflammation and promotes hippocampal neurogenesis through PPARgamma involvement. PLoS One. 2011;6(12):e28668. doi: 10.1371/journal.pone.0028668. Epub 2011 Dec 5. PMID 22163051
- [Background] Campos AC, Moreira FA, Gomes FV, Del Bel EA, Guimaraes FS. Multiple mechanisms involved in the large-spectrum therapeutic potential of cannabidiol in psychiatric disorders. Philos Trans R Soc Lond B Biol Sci. 2012 Dec 5;367(1607):3364-78. doi: 10.1098/rstb.2011.0389. PMID 23108553
- [Background] Costa B, Giagnoni G, Franke C, Trovato AE, Colleoni M. Vanilloid TRPV1 receptor mediates the antihyperalgesic effect of the nonpsychoactive cannabinoid, cannabidiol, in a rat model of acute inflammation. Br J Pharmacol. 2004 Sep;143(2):247-50. doi: 10.1038/sj.bjp.0705920. Epub 2004 Aug 16. PMID 15313881
- [Background] Bisogno T, Hanus L, De Petrocellis L, Tchilibon S, Ponde DE, Brandi I, Moriello AS, Davis JB, Mechoulam R, Di Marzo V. Molecular targets for cannabidiol and its synthetic analogues: effect on vanilloid VR1 receptors and on the cellular uptake and enzymatic hydrolysis of anandamide. Br J Pharmacol. 2001 Oct;134(4):845-52. doi: 10.1038/sj.bjp.0704327. PMID 11606325
- [Background] Walitt B, Klose P, Fitzcharles MA, Phillips T, Hauser W. Cannabinoids for fibromyalgia. Cochrane Database Syst Rev. 2016 Jul 18;7(7):CD011694. doi: 10.1002/14651858.CD011694.pub2. PMID 27428009
- [Background] Blumenthal DE, Malemud CJ. Recent strategies for drug development in fibromyalgia syndrome. Expert Rev Neurother. 2016 Dec;16(12):1407-1411. doi: 10.1080/14737175.2016.1207531. Epub 2016 Jul 14. PMID 27362466
- [Background] Babson KA, Sottile J, Morabito D. Cannabis, Cannabinoids, and Sleep: a Review of the Literature. Curr Psychiatry Rep. 2017 Apr;19(4):23. doi: 10.1007/s11920-017-0775-9. PMID 28349316
- [Background] Clark AJ, Lynch ME, Ware M, Beaulieu P, McGilveray IJ, Gourlay D. Guidelines for the use of cannabinoid compounds in chronic pain. Pain Res Manag. 2005 Autumn;10 Suppl A:44A-6A. doi: 10.1155/2005/894781. PMID 16237482